CLINICAL TRIAL: NCT06630260
Title: A Phase 1/2 Trial of the Doublet Combination of Avutometinib and Defactinib and as a Triplet in Combination With Temozolomide in Patients With High Grade Malignant Brain Tumours Within the 5G Platform
Brief Title: 5G-RUBY: Avutometinib and Defactinib in Malignant Brain Tumours
Acronym: 5G-RUBY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Minderoo Foundation (Unknown); Verastem, Inc. (Industry); Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Research UK (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5812
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme (GBM); Glioblastoma Multiform (Grade IV Astrocytoma); Diffuse Hemispheric Glioma, H3 G34-Mutant; Malignant Primary Gliomas
MeSH Terms: conditions — Glioblastoma | interventions — defactinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): The Phase 1b will evaluate the safety and tolerability of combination of avutometinib and defactinib and determine its preliminary antitumour activity when administered at the recommended Phase 2 dose (RP2D) in patients with molecularly defined malignant brain tumours.
  Interventions: Drug: Avutometinib; Drug: Defactinib
- Phase 2 (Experimental): The Phase 2 part of the study will determine the antitumour activity of investigational agents administered at the RP2D in patients with molecularly defined malignant brain tumours. Avutometinib and defactinib may be administered in combination with temozolomide (TMZ).
  Interventions: Drug: Avutometinib; Drug: Defactinib; Drug: Temozolomide

INTERVENTIONS:
Drug: Avutometinib — Supplied as 0.8mg capsules.
  Other Names: VS-6766
Drug: Defactinib — Supplied as 200mg tablets.
Drug: Temozolomide — Temozolomide will be supplied as 5, 20, 100, 140, 180 or 250 mg hard capsules.
  Other Names: Temodal
  Arms: Phase 2

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of avutometinib and defactinib and to determine the preliminary antitumour activity of avutometinib and defactinib administered at the recommended Phase 2 dose (RP2D). In the Phase 1b of this study parallel biomarker defined arms will be opened, initially in the relapsed GMB setting, enrolling 12 patients onto each arm. These patients will be treated with avutometinib and defactinib double therapy. Avutometinib will be administered orally at 3.2mg twice a week (e.g., on Monday / Thursday or Tuesday / Friday) with or without a meal. The total weekly dose of avutometinib is 6.4mg. Defactinib will be administered orally, at 200mg, twice a day within 30 min after a meal. The total daily dose of defactinib is 400mg.

Once a treatment in any biomarker arm has met the "GO" decision (≥3 successes/12 patients) for relapsed GBM in Phase 1b, that arm can progress to Phase 2. The primary objective of Phase 2 is to determine the antitumour activity of investigational agents administered at the RP2D in patients with molecularly defined malignant brain tumours.

DETAILED DESCRIPTION:
The clinical trial will be divided into two parts: Phase 1b (proof of concept of hypothesis-driven biomarker-guided therapies) and Phase 2 (preliminary efficacy testing).

This is a study within Minderoo 5G: A Next Generation AGile Genomically Guided Glioma Modular Platform for proof-of-concept molecular hypothesis testing in patients with high grade malignant brain tumours.

5G-RUBY is a Bayesian multi-centre, multi-arm, open-label, adaptive, seamless Phase 1/2 trial of doublet combination of avutometinib and defactinib and triplet combination with temozolomide for patients with malignant brain tumours.

5G-RUBY will recruit patients with glioblastoma (GBM) into two molecularly-defined biomarker arms of patients who have tumours that harbour:

* Hyperactivating BRAF mutations or fusions predicted to be pathogenic by COSMIC
* NF1 loss

Each biomarker arm, within Phase 1, will have robust GO/ADAPT decision points, reviewed by the Safety Review Committee (SRC) to allow for both agility and clear direction for next steps. A 2-stage Bayesian adaptive design will be performed to assess preliminary efficacy.

In the Phase 1b of this study parallel biomarker defined arms will be opened, initially in the relapsed GMB setting, enrolling 12 patients onto each arm. These patients will be treated with avutometinib with a total weekly dose of 6.4mg, and defactinib with a total daily dose of 400mg.

Phase 2 efficacy testing will be undertaken in the front line adjuvant MRD setting. This can be either as double combination or in triple combination with temozolomide (concomitantly, or sequentially) depending on emerging data. Further details will be provided at once the SRC has assessed data from Phase 1 and formally opened Phase 2.

ELIGIBILITY:
Inclusion Criteria for Phase 1b:

1. Patients with histologically confirmed advanced WHO Stage IV glioblastoma (per fourth edition 2016). Per the new 2021 fifth edition of WHO Classification of Tumours of the Central Nervous System, this will include:

   * Glioblastoma, IDH-wildtype Grade 4
   * Astrocytoma, IDH-mutant, Grade 4 (lower Grade 2/3 are not included)
   * Diffuse hemispheric glioma, H3 G34 mutant Grade 4

   Patients with any other CNS tumours will only be eligible for defined Phase 2 biomarker arms once a Phase 1b GO decision has been met. Specific eligibility criteria for these tumours will be defined following an amendment.
2. Patients for Phase 1 will need to have consented to the Minderoo Precision Brain Tumour Programme and have available whole genome, and transcriptome data available.
3. Patients for the relapsed cohorts will be eligible at first relapse following completion of optimal surgery, and Stupp based adjuvant chemo-radiotherapy (or equivalent). They will need to have measurable disease per RANO or evaluable disease.
4. Patients for the front line minimal residual disease (mrd) cohort will be eligible following completion of optimal surgery and Stupp based adjuvant chemoradiotherapy as long as they meet all other inclusion/exclusion criteria.
5. 16 years or over
6. Life expectancy of at least 12 weeks.
7. World Health Organisation (WHO) performance status of 0-1
8. Neurologically stable (e.g., without a progression of neurological symptoms or requiring escalating doses of systemic steroid therapy within the last week)
9. Written (signed or dated) informed consent and be capable of co-operating with treatment and follow up
10. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week prior to the first dose of either IMP

    Haemoglobin (Hb): ≥ 9.0 g/dL; Absolute neutrophil count: ≥1.5 x 10^9/L; Platelet count: ≥100 x 10^9/L; Coagulation: INR <1.5 and APTT <1.5x if not anticoagulated, INR stable > 7 days within intended therapeutic range if anticoagulated; Bilirubin: Within institution normal ranges; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): <3 x ULN; Albumin: ≥ 28 g/dL; Creatinine: <1.5 x ULN; Sodium: ≥130 mmol/L; Potassium, Calcium, Magnesium, phosphate: Within institution normal ranges (replacement is permitted); Urinary protein: < 1+ on dipstick.
11. Female patients with reproductive potential must have a negative serum pregnancy test within 14 days prior to start of trial.
12. Men and women of childbearing potential must agree to comply with the use of a highly effective method of contraception to avoid impregnating a partner or becoming pregnant, respectively, during the study, and for at least 150 days after the last dose of either investigational drug.

Exclusion Criteria for Phase 1b:

1. Receipt of treatment before the first dose of study drug (Cycle 1 Day 1) within an interval shorter than the following, as applicable:

   * Cytotoxic chemotherapy during the prior 2 weeks or 6 weeks for nitrosoureas
   * Bevacizumab during the prior 6 weeks
   * Five half-lives of any small molecule investigational or licensed medicinal product.
2. Prior immune checkpoint inhibitor therapy or vaccine therapy is not permitted. Prior use of any other immune-modulatory investigational agent must be discussed with sponsor team and CI. Prior use of BRAF or MEK inhibitors is not permitted.
3. Ongoing Grade 2 or greater toxicities from pre-existing conditions or from previous treatments.
4. Patients with carcinomatous meningitis, leptomeningeal spread of tumour, spread of tumour to the brain stem or spinal cord.
5. Has evidence of recent intratumoural or peritumoural haemorrhage on baseline MRI. Patients with radiological findings that are stable on at least 2 consecutive MRI scans at least 3 weeks apart will be eligible.
6. History of clinically relevant bleeding disorders, including significant GI bleeding within last 6 months.
7. History of arterial thromboembolism.
8. Recent (within 3 months) deep vein thrombosis or pulmonary embolism or another significant thromboembolism. Venous port of catheter thrombosis or superficial thrombosis are not considered significant. Patients with prior thrombosis (> 3 months ago) on stable anticoagulation are permitted to be enrolled. Patients on Warfarin will need to be converted onto low-molecular weight-based heparin therapy.
9. History of clinically significant cardiac disorders:

   * Myocardial infarction, or New York Heart Association Class II to IV congestive heart failure, within 6 months of the first dose of study drug
   * Concurrent and clinically significant abnormalities on ECG at Screening, including a corrected QT interval (QTcF >460ms).
10. History of malabsorption syndrome or other conditions that may interfere with enteral absorption. Patients with a history of or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis). Patients with acute or chronic pancreatitis. History of gastrointestinal perforation or fistulae. Patients with known Gilbert's syndrome will be excluded from this study.
11. Concurrent ocular disorders:

    1. Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes
    2. Patient with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    3. Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
12. Has urine protein > 1g/24 hours. Participants with >1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria.
13. Has significant lung disease including pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, active tuberculosis, or history of opportunistic infections (including PCP or CMV pneumonia).
14. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
15. Steroid requirement for neurological symptom control of > 3mg Dexamethasone per day (patients will allowed to enrol if they have been on a stable dose of steroids of equivalent or less than 3mg Dexamethasone for at least 5 days prior to Day 1 of Cycle 1).
16. Has received a live vaccine within 30 days of planned start of study therapy. Note: inactive vaccines including COVID vaccines are allowed prior to 1 week of Day 1 of Cycle 1).
17. Current active concurrent malignancy. Cancer survivors who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease recurrence for three years or more and are deemed at negligible risk of recurrence will be eligible.
18. Is a participant or plans to participate on another interventional clinical trial while taking part in this Phase 1 study. Participation in an observational trial would be acceptable.
19. Exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with study interventions within 14 days prior to the first dose of study intervention and during the course of therapy, including:

    1. Strong CYP3A4 inhibitors or inducers, due to potential drug-drug interactions with both avutometinib and defactinib.
    2. Strong CYP2C9 inhibitors or inducers, due to potential drug-drug interactions with defactinib. Not applicable if and when patients randomized to avutometinib monotherapy.
    3. Strong P-glycoprotein (P-gp) inhibitors or inducers, due to potential drug-drug interactions with both avutometinib and defactinib.
    4. Strong breast cancer resistance protein (BCRP) inhibitors or inducers, due to potential drug-drug interactions with avutometinib.
20. Major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or palliative radiotherapy within 1 week of the first dose of defactinib.
21. Any other condition which in the investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - To evaluate the safety and tolerability of investigational agent in patients with malignant brain tumours | 12 months
  To identify the incidence, nature and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Phase 1b - To determine the preliminary antitumour activity of the investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 12 months
  Antitumour activity will be defined on the basis of the following outcomes. If any of the following occur, patients will be considered to have clinically benefitted:
  For relapsed GBM:
  Achievement of overall response of CR or PR per Response Assessment in Neuro-Oncology (RANO) within 6 months or Free of disease progression or death at 6 months
  For front line unmethylated GBM (MRD):
  • Progression-free survival (PFS)
Phase 2 - To determine the antitumour activity of investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 9 months
  Antitumour activity will be defined on the basis of the following outcomes:
  Progression-free survival (PFS), defined as the time from enrolment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RANO Overall survival (OS), defined as the time from enrolment to death from any cause

SECONDARY OUTCOMES:
Phase 1b - To identify molecular determinants of response and antitumour activity of the investigational agent in patients with molecularly selected brain tumours | 12 months
  Determine biomarkers of response, including but not limited to genomic, transcriptomic or immunological signatures from responders and non-responders.
Phase 2 - To identify molecular determinants of response and antitumour activity of the investigational agent in patients with molecularly selected brain tumours | 9 months
  Determine biomarkers of response, including but not limited to genomic, transcriptomic or immunological signatures from responders and non-responders from archival tumour samples
Phase 2 - To assess changes in Quality of Life over time | 9 months
  Global changes over time in health-related quality of life (HRQOL) as assessed by the EORTC QLQ C30 and EORTC QLQ BN20 (Baseline, end of C1, C3D1)
Phase 2 - To assess safety and tolerability of combination with TMZ when given as standard of care maintenance therapy | 9 months
  To identify the incidence, nature and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Phase 2 - To assess changes in Quality of Life over time | 9 months
  PFS6, defined as the percentage of patients who remained free of disease progression 6 months from study enrolment
Phase 2 - To assess changes in Quality of Life over time | 9 months
  OS12, defined as the percentage of patients who remained free of death at 12 months from study enrolment

OTHER OUTCOMES:
Exploratory objective - To determine mechanisms of resistance to the investigational agent in patients with malignant brain tumours | 12 months
  Correlate antitumour activity of the investigational agent with the detection of putative predictive biomarkers of response and resistance in archival tumours, patient derived cells lines and plasma samples banked as part of the Minderoo Precision Brain Tumour Programme.
Exploratory objective - To assess putative predictive biomarkers of the investigational agent in patients with malignant brain tumours | 12 months
  Correlate treatment response with co-segregating mutational landscapes and identify mechanism of precision drug resistance e.g., on target vs off target, on pathway.
Exploratory objective - To identify putative precision therapy combinations with the potential for additive benefit | 12 months
  Plan rational combination therapies based on these results.

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MD, PhD, Study Director — National Health Service, UK
Locations (3):
- United Kingdom (3):
  - Cambridge University Hospitals, Cambridge
  - The Royal Marsden Hospital - Drug Development Unit, Sutton
  - The Royal Marsden Hospital - Neuro-Oncology Unit, Sutton

IPD SHARING:
Plan to Share IPD: Undecided